CLINICAL TRIAL: NCT03572413
Title: The Effectiveness of Low Pressure Pneumoperitoneum During Laparoscopic Colorectal Surgery in Preserving Innate Immune Homeostasis by Reducing Peritoneal Mesothelial Cell Injury.
Brief Title: The Effect of Low Pressure Pneumoperitoneum During Laparoscopic Colorectal Surgery on Innate Immune Homeostasis.
Acronym: RECOVER-PLUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL65290.091.18 substudy
Record Dates: First submitted 2018-06-18; First posted 2018-06-28 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-03

CONDITIONS: Pneumoperitoneum; Neuromuscular Blockade; Surgery; Immune Suppression
Keywords: Laparoscopic surgery; Deep neuromuscular block; Low pressure pneumoperitoneum; Postoperative immune suppression
MeSH Terms: conditions — Pneumoperitoneum | interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low pressure PNP, deep NMB (Experimental): Low pressure pneumoperitoneum of 8 mmHg with deep neuromuscular block (post tetanic count of 1-2) reached by titration with continuous infusion of Rocuronium bromide.
  Interventions: Procedure: Low pressure pneumoperitoneum; Drug: Rocuronium bromide
- Normal pressure PNP, moderate NMB (Active Comparator): Normal pressure pneumoperitoneum of 12 mmHg with moderate neuromuscular block (TOF count of 1-2) reached by titration with bolus or continuous infusion of a low dose of Rocuronium bromide.
  Interventions: Drug: Rocuronium bromide

INTERVENTIONS:
Procedure: Low pressure pneumoperitoneum — Lowering intra-abdominal pressure during laparoscopic surgery
  Other Names: Low intra-abdominal pressure
  Arms: Low pressure PNP, deep NMB
Drug: Rocuronium bromide — Deep (PTC 1-2) versus moderate (TOF count 1-2) neuromuscular block
  Other Names: Deep muscle relaxation

SUMMARY:
Substudy of the RECOVER trial (a randomised controlled trial comparing the effect of low pressure pneumoperitoneum with deep neuromuscular block versus normal pressure pneumoperitoneum with moderate neuromuscular block during laparoscopic colorectal surgery on early quality of recovery) investigating innate immune homeostasis after laparoscopic colorectal surgery.

DETAILED DESCRIPTION:
Rationale: increased intra-abdominal pressure can cause peritoneal mesothelial cell injury either directly or by compression of the capillary vessels, causing a variable degree of ischemia reperfusion injury. The immune system can identify damage to host cells by recognising Danger-Associated Molecular Patterns (DAMPs) that are released upon cell death in an uncontrolled fashion, such as during surgical trauma. DAMPs elicit an immune response similar to the response to invading pathogens and induce an anti-inflammatory immune response strongly related to postoperative recovery, infectious complications and mortality. Low pressure PNP is associated with lower levels of serum pro- and anti-inflammatory cytokines and better preservation of innate immune function.

Objective: to establish the relationship between the use of low pressure pneumoperitoneum with deep neuromuscular blockade and innate immune function after laparoscopic colorectal surgery.

Study design: a multi-center, blinded, randomized controlled clinical trial.

Study population: adult individuals scheduled for laparoscopic colorectal surgery with a primary colonic anastomosis.

Intervention: participants will be randomly assigned in a 1:1 fashion to either the experimental group (group A): low pressure PNP (8 mmHg) with deep NMB (PTC 1-2) or the control group (group B): normal pressure PNP (12 mmHg) with moderate NMB (TOF count 1-2).

Primary endpoint: mononuclear cell responsiveness ex-vivo as reflected by TNFα release upon LPS stimulation.

Secondary endpoints: mononuclear cell responsiveness ex-vivo as reflected by IL-6, IL-10 and IL-1beta release upon LPS stimulation. Peritoneal mesothelial hypoxia as reflected by peritoneal HIF1α mRNA expression, histological peritoneal mesothelial cell injury and plasma levels of DAMPs and cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for laparoscopic colorectal surgery with a primary anastomosis
* Obtained informed consent
* Age over 18 years

Exclusion Criteria:

* Insufficient control of the Dutch language to read the patient information and to fill out the questionnaires
* Primary colostomy
* Neo-adjuvant chemotherapy
* Chronic use of analgesics or psychotropic drugs
* Use of NSAIDs shorter than 5 days before surgery
* Known or suspected allergy to rocuronium of sugammadex
* Neuromuscular disease
* Indication for rapid sequence induction
* Severe liver- or renal disease (creatinine clearance <30ml/min)
* BMI >35 kg/m²
* Deficiency of vitamin K dependent clotting factors or coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Mononuclear cell responsiveness ex vivo | Before surgery, 24 and 72 hours after surgery
  TNFalpha release upon LPS stimulation

SECONDARY OUTCOMES:
Mononuclear cell responsiveness ex-vivo | Before surgery, 24 and 72 hours after surgery
  IL-6, IL-10 and IL-1beta release upon LPS stimulation
Serum DAMPs and cytokines | Before surgery, at the end of surgery and 24 hours after surgery
  Danger associated molecular patterns, TNFalpha, IL-6 and IL-10
HLA-DR mRNA expression | Before surgery, 24 and 72 hours after surgery
  MHC-II antigen presenting immune receptor
Peritoneal histology and HIF1alpha expression | At the start and end of surgery
  Histology and HIF1alpha mRNA expression of a peritoneal biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Kim I Albers, MD, Principal Investigator — Radboud University Medical Center; Michiel C Warlé, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Canisius Wilhelmina Hospital, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No